CLINICAL TRIAL: NCT06607380
Title: A Randomized, Open-Label, Parallel-Design Pharmacokinetic and Pharmacodynamic Interaction Study of TNM002 and Adsorbed Tetanus Vaccine Administered Alone and Simultaneously Administered in Chinese Healthy Subjects
Brief Title: A Randomized, Open-Label, Parallel-Design Pharmacokinetic and Pharmacodynamic Interaction Study of TNM002 and Adsorbed Tetanus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNM002-P1-CH02
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): TNM002
  Interventions: Biological: TNM002
- Group 2 (Active Comparator): Adsorbed tetanus vaccine
  Interventions: Biological: Adsorbed tetanus vaccine
- Group 3 (Experimental): TNM002 + adsorbed tetanus vaccine
  Interventions: Biological: TNM002 + adsorbed tetanus vaccine

INTERVENTIONS:
Biological: TNM002 — A single intramuscular (IM) gluteal injection
  Arms: Group 1
Biological: Adsorbed tetanus vaccine — A single IM deltoid injection
  Arms: Group 2
Biological: TNM002 + adsorbed tetanus vaccine — A single IM gluteal injection+ a single IM deltoid injection
  Arms: Group 3

SUMMARY:
This study is designed as a randomized, open-label, parallel-design study to evaluate the effect of TNM002 simultaneously administered with adsorbed tetanus vaccine on the PK, PD and immunogenicity properties of TNM002 and on the PD properties of the adsorbed tetanus vaccine, and to evaluate the safety and tolerability of TNM002 administered alone and simultaneously administered with adsorbed tetanus vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 18-55 years of age (inclusive) at enrollment;
2. Subjects who voluntarily provide signed written ICF;
3. Subjects who are able to well communicate with investigator as well as understand and adhere to the requirements of this study;

Exclusion Criteria:

1. Previous history of gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncologic, respiratory, immunological, cardiovascular and cerebrovascular diseases, which, as judged by the investigator, may affect the safety of the patient or may affect the PK, PD or immunogenicity assessment of this study;
2. Exposure to tetanus vaccines or vaccines containing antigenic components of tetanus toxoid within the past 10 years;
3. Exposure to tetanus immunoglobulin, receipt of blood transfusion or use of blood products within the past 6 months prior to screening;
4. History or family history of neurologic symptoms such as convulsions, epilepsy, encephalopathy and psychosis;
5. Subjects with thrombopenia or other coagulation disorders, or bleeding constitution or bleeding time prolongation, which may cause contraindications to IM injection;
6. Subjects with any acute illness requiring systemic antibiotics or antiviral therapy within 7 days prior to screening. Subjects with fever within 3 days prior to screening;
7. Receipt of immunosuppressants or immunopotentiators, other than inhaled or topical immunosuppressants within 3 months prior to dosing;
8. Allergy to the investigational product or its excipients, or have a history of allergy to vaccines or human immunoglobulin products or other therapeutic monoclonal antibodies (mAbs);
9. History of surgery within 3 months prior to screening, or planned surgery during the study;
10. Known or suspected history of drug abuse within 5 years prior to screening, or with positive urine drug abuse screening result; or a previous history of drug addiction;
11. Participation in other clinical studies with the investigational drugs or devices within 3 months or within 5 times the half-life of the specific drugs/biological products prior to dosing, except for observational, non-interventional clinical studies;
12. Use of any other drug, including over-the-counter medications and Chinese herbal medicines within 14 days prior to dosing ;
13. Exposure to other vaccines within 1 month prior to dosing, or plan to receive live vaccines within 3 months after dosing;
14. Pregnant or lactating women;

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-13 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of TNM002, area under the plasma concentration-time curve from time 0 to the last quantifiable time point post-dose (AUC0-last) | Up to Day 106
Percentage of subjects with an increase of serum TNM002-specific anti-tetanus neutralizing antibody titers (ΔTiters) ≥ 0.01 IU/mL from baseline at 24 hours after immunization | Up to 24 hours after administration
Percentage of subjects with serum anti-tetanus antibody titers ≥ 0.1 IU/mL on 28 days after immunization | Up to 28 days after administration

SECONDARY OUTCOMES:
Time to maximum serum TNM002 concentration (Tmax), elimination half-life (t1/2), and if data permit, apparent clearance (CL/F) and apparent volume of distribution (Vz/F) after immunization | Up to Day 106
Percentage of subjects with anti-tetanus neutralizing antibody ΔTiters ≥ 0.01 IU/mL at post-dose time points other than 24 hours after immunization | Up to Day 106
Serum TNM002-specific anti-tetanus neutralizing antibody titer and ΔTiters at each post-dose time point after immunization | Up to Day 106
Percentage of subjects with anti-tetanus antibody titer ≥ 0.1 IU/mL at post-dose time points other than 28 days after immunization | Up to Day 106
Percentage of subjects with serum anti-tetanus antibody titer ≥ 1.0 IU/mL at each post-dose time point after immunization | Up to Day 106
Serum anti-tetanus antibody titers, and fold increases from baseline at each post-dose time point | Up to Day 106
Adverse events (AEs), safety laboratory test, 12-lead electrocardiogram (ECG), physical examination, and vital signs | Up to Day 106
Percentage of subjects with positive anti-TNM002 antibody (ADA) in serum. | Up to Day 106

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Doctor, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification.
Supporting Information: Study Protocol
Time Frame: Starting 6 months and ending 5 years following article publication.
Access Criteria: Academics who provide a methodologically sound proposal. The leading clinical site and sponsor will review the request.